CLINICAL TRIAL: NCT05660746
Title: Precise Infliximab Exposure and Pharmacodynamic Control to Achieve Deep Remission in Pediatric Crohn's Disease
Brief Title: Precise Infliximab Exposure and Pharmacodynamic Control
Acronym: REMODEL-CD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0071; R01DK132408-01 (NIH)
Record Dates: First submitted 2022-11-29; First posted 2022-12-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease
Keywords: Crohn's
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Intervention Model Description: Patients newly diagnosed with Crohn's disease (ages 6-22 years inclusive) within the last 90 days AND starting infliximab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Conventional dosing (Active Comparator): Induction Phase: 5-7.5 mg/kg at 0, 2, and 6 weeks. Maintenance Phase : 5-10 mg/kg at every 4-8 weeks based on results of drug concentration monitoring for a flat target of 5-10 μg/mL.
  Interventions: Drug: Infliximab
- Precision dosing (Experimental): Induction: 5-12.5 mg/kg at 0, 2, and 6 weeks to target a week6 concentration of 18-24 μg/mL with dosing support provided by the RoadMABTM clinical decision support tool. Maintenance: 5-15 mg/kg every 4-8 weeks to achieve apriori pharmacokinetic and pharmacodynamic targets (CRP, disease activity scores and fecal calprotectin) with dosing support provided by the RoadMABTM clinical decision support tool.
  Interventions: Device: RoadMAB; Drug: Infliximab

INTERVENTIONS:
Device: RoadMAB — The RoadMAB Dashboard is a real-time decision support system that incorporates PK model-informed Bayesian estimation to provide precision dosing at the point of care.
  Arms: Precision dosing
Drug: Infliximab — Conventional dosing. Induction: 5-7.5 mg/kg at 0, 2, and 6 weeks. Maintenance: 5-10 mg/kg at every 4-8 weeks based on results of drug concentration monitoring for a flat target of 5-10 μg/mL.
  Precision dosing. Induction: 5-12.5 mg/kg at 0, 2, and 6 weeks to target a week6 concentration of 18-24 μg/mL with dosing support provided by the RoadMABTM clinical decision support tool. Maintenance: 5-15 mg/kg every 4-8 weeks to achieve apriori pharmacokinetic and pharmacodynamic targets (CRP, disease activity scores and fecal calprotectin) with dosing support provided by the RoadMABTM clinical decision support tool.
  Other Names: Avsola; Inflectra; Ixifi; Remicade; Renflexis

SUMMARY:
Approximately 3 million people in the United States are living with inflammatory bowel disease, which includes Crohn's Disease (CD). There are limited treatment options approved for use in children and adults with Crohn's disease. Physicians need better ways to inform decisions on treatment.

The main reason for this research study is to determine if a computer program that calculates an individualized dose based on a patient's blood testing results (precision dosing) can better achieve the best possible response to infliximab compared to standard dosing (conventional dosing).

DETAILED DESCRIPTION:
This is an open-label, cluster randomized clinical trial to test whether precision infliximab dosing with a targeted concentration intervention is superior in achieving deep remission (endoscopic healing and clinical remission) compared to patients receiving conventional infliximab dosing.

With recognition that CD patients who achieve the "target" of deep remission with anti-TNF dose optimizations following pharmacodynamic monitoring had a significant reduction in CD-related adverse events, our central hypothesis is precision dosing with infliximab during induction and maintenance will achieve superior rates of deep remission vs. conventional care (control arm)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from the patient (≥18 years old) or from parent/legal guardian if patient is <18 years old
2. Written informed assent from patient when age appropriate
3. Diagnosis of Crohn's disease within the last 90 days (luminal-only or luminal with a perianal fistula or abscess treated with antibiotics for at least 7 days)
4. ≥6 years to ≤22 years of age, anti-TNF naïve and starting infliximab
5. Clinical activity and luminal inflammation, defined by both (1) and (2)

   * (1) PCDAI≥10 (<18 years old) or CDAI ≥150 (≥18 years old) in last 60 days before the decision to start infliximab
   * (2) SES-CD>6, or SES-CD>3 for isolated ileal disease (or a report of large intestinal ulcerations)* within the last 60 days or a fecal calprotectin >250 μg/g within last 75 days prior to screening
6. C-reactive protein >1.0 mg/dL in last 30 days and/or fecal calprotectin >250 μg/g within last 75 days prior to screening
7. Negative TB (tuberculosis) interferon-gamma release test and a negative urine pregnancy test for female patients (if menstruation has started)

Exclusion Criteria:

1. Diagnosis of ulcerative colitis or inflammatory bowel disease-unspecified
2. Prior use of anti-TNF therapy (infliximab, adalimumab, certolizumab pegol, or golimumab)
3. Internal (abdominal/pelvic) penetrating fistula(e) in last 180 days
4. Intra-abdominal abscess/phlegmon/inflammatory mass in the last 180 days
5. Active perianal abscess (receiving oral antibiotics for <7 days)
6. Intestinal stricture (luminal narrowing with pre-stenotic dilation >3 cm) and surgery planned in the next 90 days
7. Have tested positive for Clostridium difficile toxin (stool assay) or other intestinal pathogens within 14 days of screening unless a repeat examination is negative and there are no signs of ongoing infection with that pathogen.
8. Current hospitalization for complications of severe Crohn's disease
9. Planned use of methotrexate or 6-mercaptopurine (azathioprine) during the induction (first 3 doses of infliximab) phase
10. Current ileostomy, colostomy, ileoanal pouch, and/or previous extensive small bowel resection (>35 cm) or any CD surgery planned within the next 90 days
11. History of autoimmune hepatitis, primary sclerosing cholangitis, thyroiditis, or juvenile idiopathic arthritis
12. Treatment with another investigational drug in the last four weeks
13. History of malignancy (including lymphoma or leukemia)
14. Currently receiving treatment for histoplasmosis
15. History of TB, human immunodeficiency virus (HIV), an immunodeficiency syndrome, a central nervous system demyelinating disease, history of heart failure or receiving intravenous antibiotics in last 14 days for any infection
16. Currently pregnant, breast feeding or plans to become pregnant in the next 1 year
17. Inability or failure to provide informed assent/consent
18. Any developmental disabilities that would impede providing assent/consent

Ages: 6 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Deep Remission | Week 52
  Pediatric Crohn's disease activity index (PCDAI) <10 (child) or Crohn's disease activity index<150 (adult), off prednisone/budesonide for >8 weeks and Simple Endoscopic Scorer Crohn's Disease (SES-CD) SES-CD≤2

SECONDARY OUTCOMES:
Rate of Steroid-free Clinical Remission | Week 14 and Week 52
  Pediatric Crohn's disease activity index (PCDAI) <10 (child) or Crohn's disease activity index(CDAI)<150 (adult) and off prednisone/budesonide for ≥4 weeks
Rate of Clinical Response | Week 14 and Week 52
  Decrease from baseline PCDAI of at least 12.5 points & total PCDAI<30 or a PCDAI<10 (child) or a reduction of CDAI>70 from baseline or CDAI<150 (adult)
Rate of Primary Clinical Nonresponse | Week 16
  On prednisone >16 consecutive weeks from start of infliximab or a PCDAI>30 or CDAI>220 for first four infusions
Rate of Primary Biologic Nonresponse | Week 16
  Failure to improve baseline fecal calprotectin by >100 μg/g (limited to patients with a baseline fecal calprotectin >250 μg/g) or Failure to improve baseline c-reactive protein ≥0.5 mg/dL (limited to patients with a baseline c-reactive protein >1.0 mg/dL)
Rate of Sustained Steroid-free Remission | Week 22 - Week 52
  PCDAI<10 (child) or CDAI<150 (adult) at dose5 to week52 and off prednisone/budesonide from week 22-52
Rate of Steroid-free Remission -biomarker composite | Week 14 and Week 52
  PCDAI<10 (child) or CDAI<150 (adult), off prednisone/budesonide for ≥4 weeks, CRP≤0.5 mg/dL and fecal calprotectin <250 μg/g
Rate of Endoscopic Healing | Week 52
  Simple endoscopic score-Crohn's disease (SES-CD) ≤2
Rate of Complete Endoscopic Healing | Week 52
  SES-CD=0
Rate of Endoscopic Remission | Week 52
  SES-CD<4
Rate of Mucosal Healing | Week 52
  SES-CD≤2 and Ileal Global Histologic Activity Score (GHAS)/ Colon Global Histologic Activity Score (CGHAS) ≤2
PK Model Bias | Week 0 - Week 52
  Model predicted vs. actual infliximab concentration. Bias: mean predictive error (MPE)
PK Model Precision | Week 0 - Week 52
  Model predicted vs. actual infliximab concentration. Precision: root mean squared error (RMSE)
Rate of IBD related event - Fistula | Week 0 - Week 52
  Occurrence of fistula and presence of antibody to infliximab >200 ng/mL
Rate of IBD related - Hospitalization | Week 0 - Week 52
  Occurrence of Crohn's disease related hospitalization
Rate of IBD related event - Surgery | Week 0 - Week 52
  Occurrence of Crohn's disease related surgery
Rate of IBD related event - Intestinal stricture | Week 0 - Week 52
  Occurrence of Crohn's disease related intestinal stricture
Rate of IBD related event - Starting corticosteroids | Week 0 - Week 52
  Occurrence of subjects starting a corticosteroid after week20
Rate of IBD related event - Antibodies to infliximab | Week 0 - Week 52
  Occurrence of antibodies to infliximab defined as >200 ng/mL
Rate of Growth Restoration - Weight change | Week 14 - Week 52
  In Tanner stage I-III subjects: change in baseline weight (kg) by gender and age group
Rate of Growth Restoration- Height velocity | Week 14 - Week 52
  In Tanner stage I-III subjects: change in height velocity (z-score) by gender
PK of infliximab in pediatric patients | Week 0 - Week 52
  Measured infliximab clearance at baseline and at week52
Correlation between infliximab induction exposure and endoscopic remission | Exposure Week 0 - Week 14, Efficacy Week 52
  The correlation analysis to be performed for the total area under the curve (infliximab exposure, μg*h/mL from week0-week14) and patients achieving endoscopic remission. Endoscopic remission is defined as a SES-CD≤2.
Correlation between infliximab induction exposure and deep remission | Exposure Week 0 - Week 14, Efficacy Week 52
  The correlation analysis to be performed for the total area under the curve (infliximab exposure, μg*h/mL from week0-week14) and patients in deep remission. Deep remission is defined as a PCDAI<10 (child) or CDAI<150 (adult), off prednisone/budesonide for >8 weeks and a SES-CD≤2.
Patient Reported Outcome-2 (PRO2) Response | Week 6, Week 14, Week 26, Week 52
  >50% improvement in total score from baseline
Patient Reported Outcome-2 (PRO2) Remission | Week 6, Week 14, Week 26, Week 52
  Stool frequency ≤3.0 and abdominal pain ≤1.0 (from baseline)
Quality of Life & Disability -IMPACT-III score | Week 52
  Total IMPACT-III (child) score
Quality of Life & Disability - Inflammatory Bowel Disease Disk score | Week 52
  Total Inflammatory Bowel Disease Disk (without sexual function assessment) score
Quality of Life & Disability - Short Inflammatory Bowel Disease score | Week 52
  Total Short IBD Questionnaire (adult) score
Process Evaluation -Usability of Decision Support Tool | Week 0 - Week 52
  Total System Usability Scale score
Rate of Adverse events | Week 0 - Week 52
  Number of Adverse Events
Rate of Serious Adverse events | Week 0 - Week 52
  Number of Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Minar, MD,MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (11):
- United States (11):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Nemours Children's Health System-Wilmington, Wilmington, Delaware
  - Nemours Children's Health System-Jacksonville, Jacksonville, Florida
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Specialty Group, Norfolk, Virginia
  - Medical College of Wisconsin, Children's of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minar PP, Colman RJ, Zhang N, Mizuno T, Vinks AA. Precise infliximab exposure and pharmacodynamic control to achieve deep remission in paediatric Crohn's disease (REMODEL-CD): study protocol for a multicentre, open-label, pragmatic clinical trial in the USA. BMJ Open. 2024 Mar 25;14(3):e077193. doi: 10.1136/bmjopen-2023-077193. PMID 38531570